CLINICAL TRIAL: NCT01575418
Title: An Exploratory, Double-Blinded, Randomized, Pharmacokinetic and Safety Study of Three Rectally-Applied Tenofovir 1% Microbicide Gel Formulations
Brief Title: An Exploratory Rectal Safety Study of Three Tenofovir Gel Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ian McGowan (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); CONRAD (Other)
Responsible Party: Sponsor-Investigator, Ian McGowan, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: CHARM-02; 5U19AI082637 (NIH)
Record Dates: First submitted 2012-03-01; First posted 2012-04-11 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: HIV Prevention
MeSH Terms: interventions — Tenofovir; Gels; Seeds

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rectal specific formulation (RF) stage (Experimental): Each participant will receive two inpatient doses of each radiolabeled study product. The first inpatient dose of each product will be administered without coital dynamics simulation (CDS), while the second inpatient dose will be followed by a CDS procedure at 1-hour post dose with instillation of radiolabeled autologous semen. There will be a washout period of at least 11 days between each dose.
  Interventions: Drug: Rectal formulation (RF) of tenofovir 1% gel; Radiation: Radiolabeling of study drugs and semen
- Vaginal formulation (VF) stage (Active Comparator): Each participant will receive two inpatient doses of each radiolabeled study product. The first inpatient dose of each product will be administered without coital dynamics simulation (CDS), while the second inpatient dose will be followed by a CDS procedure at 1-hour post dose with instillation of radiolabeled autologous semen. There will be a washout period of at least 11 days between each dose.
  Interventions: Drug: Vaginal formulation (VF) of tenofovir 1% gel; Radiation: Radiolabeling of study drugs and semen
- Reduced glycerin vaginal formulation (RGVF) stage (Active Comparator): Each participant will receive two inpatient doses of each radiolabeled study product. The first inpatient dose of each product will be administered without coital dynamics simulation (CDS), while the second inpatient dose will be followed by a CDS procedure at 1-hour post dose with instillation of radiolabeled autologous semen. There will be a washout period of at least 11 days between each dose.
  Interventions: Drug: Reduced glycerin vaginal formulation (RGVF) of tenofovir 1% gel; Radiation: Radiolabeling of study drugs and semen

INTERVENTIONS:
Drug: Rectal formulation (RF) of tenofovir 1% gel — The RF is translucent colorless viscous gel formulation containing 1% (w/w) of tenofovir (PMPA) formulated in purified water with EDTA, glycerin, methylparaben, propylparaben, carbopol, sodium carboxy methyl cellulose, and pH adjusted to 7. The RF is close to isoosmolar with an osmolality of 479 mOsmol/kg.
  Arms: Rectal specific formulation (RF) stage
Drug: Vaginal formulation (VF) of tenofovir 1% gel — The original VF is a transparent, viscous gel formulation containing 1% (weight/ weight or w/w) of tenofovir (PMPA, 9-[(R)-2-(phosphonomethoxy)propyl]adenine monohydrate), formulated in purified water with edetate disodium, citric acid, glycerin, methylparaben, propylparaben, hydroxyethylcellulose, and pH adjusted to 4-5. This formulation has been used in all clinical trials (vaginal, penile, and rectal) of tenofovir 1% gel to date.
  Arms: Vaginal formulation (VF) stage
Drug: Reduced glycerin vaginal formulation (RGVF) of tenofovir 1% gel — Modified slightly from the original VF formulation, the RGVF has a lower glycerin content than the VF and a significantly reduced osmolality (836 or 846 versus 3111 mOsmol/kg). Lowering glycerin content lowered the viscosity, so the HEC concentration was increased by 10% (a change considered to be insignificant). The amount of parabens was increased by 10% each to improve the antimicrobical effectiveness. The RGVF formulation with 2.75% HEC was used in MTN-007 (CONRAD IND 73,382; currently enrolling), which is the only clinical study of this formulation. The RGVF formulation has since been modified to increase the viscosity.
  Arms: Reduced glycerin vaginal formulation (RGVF) stage
Radiation: Radiolabeling of study drugs and semen — Study products (i.e. the gel formulations) will be radiolabeled with 111In-DTPA, an FDA-approved radiopharmaceutical commonly used in diagnostic nuclear medicine studies. The delivered dose per gel study product will be approximately 100 microCuries (µCi) to allow sufficient visualization for the imaging period.
  Autologous whole semen collected from the participants at designated visits will be radiolabeled with a delivered dose of approximately 500 microCuries (µCi) of 99mTc-sulfur colloid, also an FDA-approved radiopharmaceutical commonly used in diagnostic nuclear studies. The study team at JHU has extensive experience administering these radiopharmaceuticals rectally. Both of these radiopharmaceuticals will be prepared and delivered by a commercial radiopharmacy and mixed by the study investigators with the respective gel and whole semen vehicles.
  The study product and autologous whole semen will be loaded into calibrated syringes with luer lock adapter for dosing.

SUMMARY:
This is a double-blinded, randomized, pharmacokinetic and safety study of 3 rectally applied tenofovir microbicide formulations: a vaginal formulation (VF), a reduced glycerin vaginal formulation (RGVF), and a rectal-specific formulation (RF). Nine HIV-negative men will be enrolled.

Each participant will receive two inpatient doses of each radiolabeled study product. The first inpatient dose of each product will be administered without coital dynamics simulation (CDS), while the second inpatient dose will be followed by a CDS procedure at 1-hour post dose with instillation of radiolabeled autologous semen. There will be a washout period of at least 11 days between each dose.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ Age of 18 at screening
2. Willing and able to communicate in English
3. Willing and able to provide written informed consent to take part in the study
4. Willing and able to provide adequate locator information
5. Understands and agrees to local STI reporting requirements
6. Biologically male
7. HIV-1 uninfected at screening according to the standard DAIDS algorithm 8. Willingness to provide semen sample on multiple occasions

9. Per participant report at screening, a history of consensual RAI at least once within the six months prior to screening 10. Willingness to perform simulated RAI with CDS device 11. Willing to abstain from RAI or any practices which include rectal insertion of any product including those used during sexual intercourse (sex toys) for 48 hours before and after inpatient dosing and willing to refrain from ejaculation for a period of 48 hours prior to each semen collection 12. Must agree to use condoms for the duration of the study 13. Must be in general good health 14. Must agree not to participate in other drug trials 15. Availability to return for all study visits, barring unforeseen circumstances

Exclusion Criteria:

1. Significant colorectal symptom(s) as determined by medical history or by participant self-report (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, history of inflammatory bowel disease, presence of symptomatic external hemorrhoids, and presence of any painful anorectal conditions that would be tender to manipulation.)
2. At screening: participant-reported symptoms and/or clinical or laboratory diagnosis of active rectal or reproductive tract infection requiring treatment per current CDC guidelines or symptomatic urinary tract infection (UTI). Infections requiring treatment include Chlamydia (CT), gonorrhea (GC), syphilis, active HSV lesions, chancroid, genital sores or ulcers, and, if clinically indicated, genital warts. Note that HSV seropositivity with no active genital lesions is not an exclusion criterion, since treatment is not required. (Note: Allow one re-screening after documented treatment (30 days) in cases where urethral GC/CT identified at screening)
3. At screening:

   * Positive for hepatitis B surface antigen
   * Calculated creatinine clearance less than 60 mL/min by the Cockcroft-Gault formula where creatinine clearance in mL/min = (140 - age in years) x (weight in kg) x (1 for male)/72 x (serum creatinine in mg/dL)
   * Alanine transaminase (ALT) and/or aspartate aminotransferase (AST) > 2.5× the site laboratory ULN
4. Known allergic reaction to methylparaben, propylparaben, sorbic acid, glycerin, glycerol, tenofovir, or other components of the test articles
5. Known HIV-infected partners
6. By participant report at enrollment, history of excessive daily alcohol use (as defined by the CDC as heavy drinking consisting of an average consumption of more than 2 drinks per day for men), frequent binge drinking or illicit drug use that includes any injection drugs, methamphetamines (crystal meth), heroin, or cocaine including crack cocaine, within the past 12 months
7. By participant report, use of any rectally-administered medications, rectally administered products containing N-9 (including condoms), any investigational products, and/or systemic immunomodulatory medications within the 4 weeks prior to the first inpatient visit and throughout study participation
8. History of recurrent urticaria
9. Participants whose whole body (EDE) radiation exposure, per the investigator's records and/or participant report, exceeds 5000mrem/year
10. Any other condition or prior therapy that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled substance abuse, or renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events and/or abnormal laboratory values Grade 2 or higher | Participants will be followed for the duration of study, an expected average of 12 weeks
  Grade 2 or higher clinical and laboratory adverse events as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, Dec 2004 and Addendum 3 (Rectal Grading Tables for Use in Microbicide Studies) will be used to assess safety.

SECONDARY OUTCOMES:
Area Under Curve (AUC) | 0.25hr, 0.5hr, 0.75hr, 1hr, 1.25hr, 1.5hr, 1.75hr, 2hr, 2.33hr, 2.66hr, 3hr, 3.5hr, 4hr, 8hr, 16hr, and 24hr post-dose at Visits 2,4,5,7,8, and 10
  Pharmacokinetics (PK) measures will be evaluated as plasma tenofovir concentrations
  Distribution/migration of product and whole semen (with and without Coital Dynamic Simulation or CDS) will be evaluated based on:
  * Distribution of product radiolabel (111Indium DTPA) within the colonic lumen
  * Distribution of whole semen radiolabel (99mTc-sulfur colloid) within the colonic lumen
  And mucosal permeability (with and without CDS) will be measured via:
  * PK in blood of product radiolabel (111Indium DTPA)
  * Urine

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hendrix, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Division of Clinical Pharmacology, Drug Development Unit, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Hiruy H, Fuchs EJ, Marzinke MA, Bakshi RP, Breakey JC, Aung WS, Manohar M, Yue C, Caffo BS, Du Y, Abebe KZ, Spiegel HM, Rohan LC, McGowan I, Hendrix CW. A Phase 1 Randomized, Blinded Comparison of the Pharmacokinetics and Colonic Distribution of Three Candidate Rectal Microbicide Formulations of Tenofovir 1% Gel with Simulated Unprotected Sex (CHARM-02). AIDS Res Hum Retroviruses. 2015 Nov;31(11):1098-108. doi: 10.1089/AID.2015.0098. Epub 2015 Aug 24. PMID 26227279